CLINICAL TRIAL: NCT01686906
Title: Mid-stromal Isolated Bowman Layer Graft Implantation to Reduce and Stabilize Advanced Keratoconus
Brief Title: Isolated Bowman Layer Graft for Reducing and Stabilizing Advanced Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Netherlands Institute for Innovative Ocular Surgery (Other)
Collaborators: Amnitrans Eyebank Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIIOS-BL-2012
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Advanced Keratoconus
Keywords: Keratoconus; Bowman layer
MeSH Terms: conditions — Keratoconus

ARMS (1):
- Bowman layer graft implantation (Experimental)
  Interventions: Procedure: Bowman layer graft implantation

INTERVENTIONS:
Procedure: Bowman layer graft implantation — For patients with progressive advanced keratoconus, a mid-stromal manual dissection is made and a donor isolated Bowman layer is positioned into the stromal pocket.

SUMMARY:
To evaluate the efficacy of mid-stromal implantation of an isolated Bowman layer graft, to reduce and stabilize ectasia in eyes with advanced keratoconus

ELIGIBILITY:
Inclusion Criteria:

•Advanced keratoconus

Exclusion Criteria:

* Further ophthalmic diseases
* History of ocular surgery
* Pregnancy, brest feeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Corneal power | 2011-2020
  Reduction and stabilizing of the corneal power after Bowman layer graft implantation

SECONDARY OUTCOMES:
Best corrected visual acuity | 2011-2020

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit RJ Melles, MD, PhD, Principal Investigator — Netherlands Institute for Innovative Ocular Surgery
Locations (1):
- Netherlands Institute for Innovative Ocular Surgery, Rotterdam, Netherlands

REFERENCES:
- [Background] van Dijk K, Liarakos VS, Parker J, Ham L, Lie JT, Groeneveld-van Beek EA, Melles GR. Bowman layer transplantation to reduce and stabilize progressive, advanced keratoconus. Ophthalmology. 2015 May;122(5):909-17. doi: 10.1016/j.ophtha.2014.12.005. Epub 2015 Jan 14. PMID 25596620
- [Background] van Dijk K, Parker J, Tong CM, Ham L, Lie JT, Groeneveld-van Beek EA, Melles GR. Midstromal isolated Bowman layer graft for reduction of advanced keratoconus: a technique to postpone penetrating or deep anterior lamellar keratoplasty. JAMA Ophthalmol. 2014 Apr 1;132(4):495-501. doi: 10.1001/jamaophthalmol.2013.5841. PMID 24557359
- [Background] Groeneveld-van Beek EA, Parker J, Lie JT, Bourgonje V, Ham L, van Dijk K, van der Wees J, Melles GR. Donor Tissue Preparation for Bowman Layer Transplantation. Cornea. 2016 Dec;35(12):1499-1502. doi: 10.1097/ICO.0000000000000905. PMID 27362885
- [Background] Parker JS, van Dijk K, Melles GR. Treatment options for advanced keratoconus: A review. Surv Ophthalmol. 2015 Sep-Oct;60(5):459-80. doi: 10.1016/j.survophthal.2015.02.004. Epub 2015 Mar 5. PMID 26077628
- [Background] van der Star L, van Dijk K, Vasiliauskaite I, Dapena I, Oellerich S, Melles GRJ. Long-Term Outcomes of Bowman Layer Inlay Transplantation for the Treatment of Progressive Keratoconus. Cornea. 2022 Sep 1;41(9):1150-1157. doi: 10.1097/ICO.0000000000002871. Epub 2021 Oct 5. PMID 34620767